CLINICAL TRIAL: NCT02373839
Title: Role of Placental Growth Factor (PlGF) in the Management of Non-Severe Preeclampsia, a Randomized Study
Brief Title: Role of Placental Growth Factor (PlGF) in the Management of Non-Severe Preeclampsia
Acronym: MAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fetal Medicine Research Center, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEIC 2013/8820
Record Dates: First submitted 2014-01-17; First posted 2015-02-27 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Pregnancy; Pre-eclampsia, Mild
MeSH Terms: conditions — Pre-Eclampsia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PlGF measurement (Other): Determination of PlGF levels. If lower than 100 pg/mL labour will be inducted at the moment of diagnosis. Otherwise standard monitoring will be done with labour induction at 37 weeks.
  Interventions: Other: Measurement of PlGF
- Controls (No Intervention): induction of labour at 37 weeks of gestation.

INTERVENTIONS:
Other: Measurement of PlGF — If lower than 100 pg/mL labour will be inducted at the moment of diagnosis. Otherwise standard monitoring will be done with labour induction at 37 weeks
  Arms: PlGF measurement

SUMMARY:
Preeclampsia is an important disease that develops during pregnancy and it is one of the main contributors to maternal and fetal complications.

The only known definitive treatment is delivery. Although delivery is always appropriate for the mother, it might not be the best for a very premature neonate.

In cases of non-severe preeclampsia there no benefit delaying delivery beyond 37 weeks. It is also well established that before 34 weeks an expectant management confers perinatal benefit with minimum amount of additional maternal risk. There is then an area of uncertainty between 37 and 37 weeks. This is why in this period it is a clinical need to select high risk patients of complications that will benefit from labor induction, and differentiate them from low risk patients that can be manage expectantly until 37 weeks.

Placental growth factor (PlGF) is an angiogenic factor that is lower in pregnant women with preeclampsia and current evidence shows that it as a predictor of adverse pregnancy outcome and requirement of delivery.

Circulating levels of PIGF at 34 weeks could help to identify those women that may benefit from labor induction and those where delivery can be delayed until 37 weeks with low risk for maternal complications.

DETAILED DESCRIPTION:
BACKGROUND

The current definition of pre-eclampsia is a new onset hypertension (>140/90mmHg) and proteinuria (>0'3g per 24 hours) after 20 weeks of gestation. Pre-eclampsia affects 3% to 8% of all pregnancies and it is a leading cause of maternal and neonatal morbidity and mortality.

It has been subclassified by clinical severity in severe and non-severe and by gestational age at the diagnosis in early and late onset pre-eclampsia (>34 weeks of gestation).

Pre-eclampsia is associated with abnormal placentation and uterine angiogenesis. Pregnant women with preeclampsia show lower circulating levels of placental growth factor (PlGF), a proangiogenic factor related to placental angiogenesis, compared with healthy pregnant women. Moreover evidence has been found regarding the role of PlGF as a predictor of adverse pregnancy outcome and requirement of delivery.

The only definitive treatment of the disease is delivery. In patients with non-severe preeclampsia between 34 and 37 weeks there is no consensus regarding the ideal time of delivery.

AIM: The aim of this study is to assess whether circulating levels of PIGF at 34 weeks could help to identify those women that may benefit from labor induction and those where delivery can be delayed until 37 weeks with low risk for maternal complications.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years
* pregnant women with non-severe preeclampsia
* gestational age between 34 and 36.5 weeks

Exclusion Criteria:

* No exclusion criteria are defined (intention-to-treat analysis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
composite of maternal complications | gestational age between 34 and 36.5 weeks
  Maternal complications as HELLP syndrome (hemolysis, elevated liver enzymes, and low platelet count), pulmonary oedema, severe hypertension, eclampsia, thromboembolic disease...
Composite of neonatal morbidity | 2 weeks
  Verma A J Epidemiol Communitary Health 2005 Score

SECONDARY OUTCOMES:
maternal risk at induction | 1 day
  according to PIERs score
Average length of maternal hospital stay | 90 days
Length of neonatal hospital stay. | 90 days
Length of maternal hospital stay | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona - Maternitat (BCNatal), Barcelona, Spain

REFERENCES:
- [Derived] Peguero A, Herraiz I, Perales A, Melchor JC, Melchor I, Marcos B, Villalain C, Martinez-Portilla R, Mazarico E, Meler E, Hernandez S, Matas I, Del Rio M, Galindo A, Figueras F. Placental growth factor testing in the management of late preterm preeclampsia without severe features: a multicenter, randomized, controlled trial. Am J Obstet Gynecol. 2021 Sep;225(3):308.e1-308.e14. doi: 10.1016/j.ajog.2021.03.044. Epub 2021 Apr 3. PMID 33823150